CLINICAL TRIAL: NCT01206218
Title: Evaluation of Customized Treatment According to BRCA1 Assessment in Patients With Advanced Gastric Cancer
Acronym: BREC-AGC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Baorui Liu, The Comprehensive Cancer Center of Drum Tower Hospital, Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREC-AGC
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Gastric Cancer
Keywords: Gastric Cancer, BRCA1
MeSH Terms: conditions — Stomach Neoplasms

ARMS (2):
- Group A (Active Comparator): FLOT Regimen
  Interventions: Drug: FLOT Regimen
- Group B (Experimental): FLO Regimen or FLOT Regimen
  Interventions: Drug: FLO Regimen or FLOT Regimen

INTERVENTIONS:
Drug: FLOT Regimen — FLOT Regimen: 5-fluorouracil, Oxaliplatin, Docetaxel
  Arms: Group A
Drug: FLO Regimen or FLOT Regimen — FLO Regimen: 5-fluorouracil, Oxaliplatin FLOT Regimen: 5-fluorouracil, Oxaliplatin, Docetaxel
  Arms: Group B

SUMMARY:
Evaluation of customized treatment according to BRCA1 assessment in patients with advanced gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Female or male aged 18 years and over
* Histologic or cytologic confirmation of advanced gastric cancer
* Stage III-IV (AJCC 7th)
* ECOG: 0-2
* Have tumor sample that can be tested for BRCA1 mRNA expression
* Negative pregnancy test for women of childbearing potential
* Neutrophile granulocyte greater than 1.5×10^9/L
* Hemoglobin greater than 10g/dL
* Platelet greater than 100×10^9/L
* Serum bilirubin not greater than 1.5x upper limit of reference range (ULRR)
* ALT or AST not greater than 1.5x ULRR
* Creatinine clearance no less than 60ml/min

Exclusion Criteria:

* Have at least another primary malignant tumor
* Active infection
* Chemotherapy with experimental drug within 3 weeks before the start of study therapy
* Women who are pregnant or breast feeding
* Weight loss greater 10% within 6 weeks before the start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 12 months

SECONDARY OUTCOMES:
Overall Survival | 12 months
Response Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Liu, MD, PHD, Principal Investigator — Drum Tower Hospital, Nanjing University Medical School